CLINICAL TRIAL: NCT01105234
Title: An Irritation Study With New Calcipotriol Ointment Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: MCO 0901 FR; 2009-017394-38 (EudraCT Number)
Record Dates: First submitted 2010-02-25; First posted 2010-04-16 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Irritation
Keywords: Healthy volunteers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcipotriol ointment (Experimental)
  Interventions: Drug: Six different calcipotriol ointment formulations, and two currently marketed topical vitamin D analogues.

INTERVENTIONS:
Drug: Six different calcipotriol ointment formulations, and two currently marketed topical vitamin D analogues.

SUMMARY:
The purpose of this trial is to compare the skin irritation potential of eight different formulations of vitamin D analogues after repeated applications on intact skin of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having understood and signed an informed consent form.
* Either sex
* Healthy subjects, 18 to 65 years of age
* Subjects with skin types I to IV according to Fitzpatrick Scale
* Subjects without erythema on test areas on the mid back skin (visual irritation score = 0) at baseline (Day 1), before randomisation.

Exclusion Criteria:

* Females who are pregnant, or who wish to become pregnant during the study, or who are breast feeding
* Any topical or systemic corticosteroids or immuno-suppressors within 3 weeks prior to randomisation
* Any other medication which may interfere with the study results, in particular topical drugs applied on the test area within 2 weeks prior to randomisation
* Any other products which may interfere with the study results, in particular emollients, creams, gels, lotions and body powders applied on the test area within 24 hours prior to randomisation
* Any systemic or cutaneous disease that may confound interpretation of the study results (e.g., atopic dermatitis, eczema, psoriasis)
* Scars, moles, sunburn, or other blemishes in the test area which may interfere with grading
* Exposure to excessive or chronic UV radiation (i.e., sunbathing, solarium, phototherapy) within 2 weeks prior to randomisation or is planned during the study period
* Known or suspected hypersensitivity to any component of the investigational products
* Participation in any other interventional clinical trial within 4 weeks prior to randomisation or during the study period, based on interview of the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Clinical scoring of the skin reaction. | 10 days
  Clinical evaluation of the irritation on 8-level scale (from score 0: no evidence of irritation, to score 7: strong reaction speading beyond the application site)

SECONDARY OUTCOMES:
Transepidermal waterloss measurements | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Facy, PhD, Study Director — LEO Pharma
Locations (1):
- LEO Pharma site, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en